CLINICAL TRIAL: NCT06796920
Title: Spinal Cord Stimulation Surgery for Improving Lower Limb Motor Dysfunction in Adrenomyeloneuropathy (AMN): A Prospective, Multicenter, Single-Arm, Self-Controlled Study.
Brief Title: Epidural Spinal Cord Stimulation for Lower-limb Impairment in Adrenomyeloneuropathy
Acronym: EPIC-AMN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other); Jingmen No.1 People's Hospital (Other); The 958th Hospital of the Chinese People's Liberation Army (Unknown)
Responsible Party: Principal Investigator, Tan Liang, Southwest hospital, Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThirdMMU-TLiang
Record Dates: First submitted 2025-01-06; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Adrenomyeloneuropathy Without Cerebral Involvement
Keywords: Genetic Diseases; Rare Diseases; Spinal Cord Stimulation; Motor Function Recovery; Multicenter Study; Adrenomyeloneuropathy
MeSH Terms: conditions — Genetic Diseases, Inborn; Rare Diseases; Adrenoleukodystrophy | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- self-controlled group (Experimental): This experiment is a single-arm trial, so there is only one group, forming a self-controlled comparison before and after the Spinal cord stimulation.
  Interventions: Procedure: Spinal cord stimulation

INTERVENTIONS:
Procedure: Spinal cord stimulation — Upon completion of the initial assessments, a lumbar spinal cord nerve stimulator and pulse generator will be implanted. Following surgery, based on the patient's recovery status, the patient will be transferred to the respective center for rehabilitation within one to two weeks. Afterward, electrical stimulation therapy will be initiated. Stimulation should be applied at least three days per week. Each day, the total stimulation time should be between 4 and 8 hours. Stimulation Modes: Continuous Stimulation: For example, if 6 hours of stimulation are prescribed, the stimulator will run uninterrupted for 6 hours. Intermittent Stimulation: For instance, a cycle of 40 seconds on and 20 seconds off. If a total of 6 hours of active stimulation is needed, the stimulator must remain on for 9 hours in total to accommodate rest intervals.The ranges for each parameter are as follows:Stimulation Frequency: 2 Hz - 2000 Hz, Pulse Width: 20 μs - 1000 μs, Stimulation Amplitude:Voltage: 0 V - 10 v

SUMMARY:
Adrenal spinal neuropathy (AMN) is a rare X-linked genetic disease caused by mutations in the ABCD1 gene, and belongs to a special type of adrenal leukodystrophy. The patient's lower limb strength is weakened, the range of motion of the ankle joint is reduced, the hip flexors are weak and affect walking, and the peripheral nerves and vibration sensation are damaged. As the condition worsens, the lower limb muscle tone changes from hyperactivity to decrease, ultimately transitioning from spastic paralysis to flaccid paralysis. At present, the treatment plan for AMN is not yet perfect, and effective therapies are urgently needed to alleviate symptoms.

Spinal cord electrical stimulation (SCS) is the implantation of a thin electrode into the epidural space of the corresponding spinal segment within the spinal canal. Then connect the electrodes to a nerve stimulator implanted subcutaneously in the iliac region, and use electrical pulses to stimulate the conduction of sensory neurons in the posterior column and posterior horn of the spinal cord for treatment, which can achieve the goal of controlling pain. In addition, SCS has also conducted research on the recovery of lower limb function in paraplegic patients and upper limb function in post-stroke hemiplegic patients, and has improved corresponding motor dysfunction to a certain extent. Spinal cord stimulation may be a potential treatment for motor dysfunction in AMN. Based on the above, this study attempts to evaluate the efficacy of SCS in treating lower limb muscle tone and movement disorders in AMN patients, and explore the potential therapeutic effects and related mechanisms of SCS on AMN.

In this study, 10 AMN patients will be recruited. After enrollment, preoperative evaluation will be conducted. After preliminary assessment of motor function, neurological evaluation, and other related examinations, lumbar spinal nerve stimulators and pulse generators were implanted in our hospital. After the implantation surgery is completed, depending on the patient's recovery status, they will be transferred to various centers for subsequent rehabilitation treatment within one to two weeks, and then turned on for treatment. Before starting up, a second corresponding inspection and evaluation will be conducted. The third and fourth corresponding inspections and evaluations will be conducted one week and four weeks after startup, respectively. The patient will be discharged 4 weeks after starting up, and then return to the hospital for the fifth and sixth corresponding examinations and evaluations at 4 weeks and 6 months after discharge. Evaluate the effectiveness and safety of SCS in improving lower limb motor dysfunction in AMN patients through statistical analysis.

DETAILED DESCRIPTION:
Adrenomyeloneuropathy (AMN) is an X-linked inherited metabolic rare disease caused by mutations in the ABCD1 gene, with an incidence rate of only 1 in 50,000. Currently, it is regarded as a special type of adrenoleukodystrophy (ALD), and AMN is the most dominant disease subtype affecting adult patients. Due to the special phenomenon of skewed X-inactivation, female heterozygotes may also have spinal cord neuropathy. Such mutations can lead to the accumulation of very long chain fatty acids (VLCFA) in the blood and organs, mainly resulting in demyelination of the central nervous system and lesions in the adrenal cortex. As the disease progresses, the strength of the lower limbs and the passive range of motion of the ankle joints of patients will gradually decline. The deterioration of hip flexor muscle weakness is closely associated with a slower walking speed and an increased degree of disability. Most patients will also experience peripheral nerve involvement and impairment of vibration sensation. Hypertonia of the lower limbs will gradually develop into a decline in both muscle strength and muscle tone, and finally progress from spastic paralysis to flaccid paralysis. However, the current commonly used treatment regimens for AMN still have deficiencies, and it is necessary to seek effective treatment methods to alleviate patients' symptoms and improve their quality of life.

Spinal Cord Stimulation (SCS) involves implanting a thin electrode (either strip-shaped or needle-shaped) into the epidural space within the spinal canal at the corresponding spinal segments, adjacent to the posterior columns of the spinal cord. The electrode is then connected to a nerve stimulator implanted subcutaneously in the iliac region, and electrical pulses are used to stimulate the conduction of the posterior columns of the spinal cord and the sensory neurons in the posterior horns for treatment purposes. This blocks the transmission of pain signals from the spinal cord to the brain, preventing them from reaching the cerebral cortex, thereby achieving the goal of pain control. Previous studies have demonstrated that, in addition to having significant therapeutic effects in analgesia, SCS has also been investigated in aspects such as the recovery of lower limb function in paraplegia and the recovery of upper limb function in hemiplegia after stroke, and it has improved the corresponding motor dysfunctions to a certain extent. For the problem of motor dysfunction in AMN, there is currently no good treatment method, and spinal cord stimulation may serve as a potential treatment approach. Based on the above, this study attempts to further explore the potential therapeutic effect and related treatment mechanisms of SCS on AMN through evaluating the efficacy of SCS in treating motor disorders of muscle tone and strength in the lower limbs of patients with AMN.

In the study, 10 patients with AMN will be recruited. After patients are enrolled in the group, preoperative evaluations will be conducted. And after the first evaluations of motor function, neurological assessment and other relevant examinations, the implantation of lumbar spinal cord nerve stimulator and pulse generator will be carried out in our hospital. After the completion of the implantation surgery, depending on the patients' recovery status, they will be transferred to each center for subsequent rehabilitation treatment within one to two weeks, and then the electrical stimulation treatment will be initiated by turning on the device. Before turning on the device, the second corresponding examinations and evaluations will be conducted. The third and fourth corresponding examinations and evaluations will be carried out one week and four weeks after turning on the device, respectively. Patients will be discharged four weeks after turning on the device, and then return to the hospital for the fifth and sixth corresponding examinations and evaluations four weeks and six months after discharge, respectively. Through the statistical analysis of self-controlled comparison before and after the trial, the efficacy and safety of SCS in improving lower limb motor dysfunction in patients with AMN will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Conforming to the diagnostic criteria of AMN, with a definite genetic testing report, and complicated by lower limb motor function disorders;
* Capable of normal communication and able to complete scale tests independently (as determined by on-site scale tests);
* Willing to participate in this study after giving informed consent;
* The muscle tone of the patient's bilateral lower extremities was elevated.

Exclusion Criteria:

* Other inherited diseases;
* Other severe central nervous system diseases;
* History of brain surgery;
* Psychiatric and psychological diseases such as depression and anxiety;
* The presence of metallic foreign bodies or prostheses (such as cardiac pacemakers, insulin pumps) in the body, claustrophobia, and other contraindications for MRI;
* Informed consent was not obtained;
* Unable to tolerate MRI-related examinations;
* Received anticoagulant, antispasmodic or antiepileptic drug therapies throughout the entire study period;
* Postoperative wound infection;
* Other motor disorders, spinal cord pathologies, fractures, osteoarthritis, amputations, scoliosis and other movement-affecting diseases.

Ages: 22 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the walking distance that patients cover in six minutes when walking as fast as possible along a straight corridor, which is a indicator for assessing the lower limb motor function.

SECONDARY OUTCOMES:
Adverse event | One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital; One year after discharge from hospital.
  Record the adverse reactions related to spinal cord stimulation (SCS), such as nerve injury, infection, hemorrhage, edema, poor wound healing, etc. These manifestations reflect the safety of spinal cord stimulation treatment.
Discomfort and pain. | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital; One year after discharge from hospital.
  This assessment is based on the fact that after each stimulus training, patients need to use the Numerical Rating Scale (NRS) to report the degree of discomfort they perceive: NRS versions 0-10 were used in this study. Use 0-10 to represent different degrees of pain: 0 represents no pain, 1-3 represents mild pain (pain does not affect sleep), 4-6 represents moderate pain (mild affects sleep), 7-9 represents severe pain (inability to fall asleep or waking up during sleep), and 10 represents severe pain.
Spinal cord and brain MRI | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the atrophy volume of each segment of the spinal cord and brain analyzed by artificial intelligence segmentation, so as to assess the progression degree of spinal cord and brain white matter injury in patients.
The degree of improvement in electrophysiological indicators of the muscles in the affected limbs | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This assessment is an objective examination of muscle electrophysiology to evaluate the recovery of the patient's motor function.
Qmax（The maximum flow rate） | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Qmax is the peak of a continuous, immediate uroflow rate numerical curve traced with a uroflowmetry device during voiding, suggesting a combination of bladder and urethral function during the subject's voiding. It is calculated in milliliters per second.
Filling bladder pressure | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Filling cystometry is a method of measuring the pressure-volume correlation of the bladder under specific media perfusion in order to understand the function of the urethra and urethra during the storage phase.
Urethral pressure | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Urethral pressure is the fluid pressure required just to open and close the urethra during urodynamics, and is an important indicator for evaluating the functional status of the urethra.
Residual urine volume | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Bladder residual urine volume is the amount of urine still remaining in the bladder after the end of urination. It is an important indicator for assessing bladder voiding function. Under normal circumstances, the residual urine volume in a healthy adult should be less than 10 milliliters. When the residual urine volume exceeds 10 milliliters, it may indicate impaired bladder voiding function.
Evaluation of erectile function (International Index of Erectile Function-5 (IIEF-5) score) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the International Index of Erectile Function (IIEF) scores. The total score of the IIEF-5 ranges from 0 to 25, and a higher score indicates that the patient has better erectile function.
Stool scoring (Wexner Incontinence Scale, Bristol Stool Scale (BSFS)) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the Wexner Incontinence Scale and the Bristol Stool Form Scale. The Wexner Incontinence Scale is a scale used to assess the severity of defecation in patients and is applicable to patients with fecal incontinence caused by various reasons. The Bristol Stool Form Scale is a classification system based on the shape of feces, which is used to evaluate the characteristics of feces and possible health problems.
Somatosensory evoked potential, visual evoked potential, auditory evoked potential, motor evoked potential. | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Evoked potentials are generated by stimulating any structures related to sensory organs, nerves, pathways or systems, resulting in measurable potential changes in the central nervous system. They can be used to assess the functional integrity of the central and peripheral nervous systems.
Motion capture (gait test) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on the range of motion of joints and spatio-temporal parameters of gait.
Short Physical Performance Battery (SPPB) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on a comprehensive score, which includes walking speed, balance tests and the chair stand test. The higher the score is, the better the physical condition will be.
Very-long-chain fatty acid (VLCFA) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  This evaluation is based on detecting the levels of very-long-chain fatty acids (VLCFAs) in plasma and cerebrospinal fluid, analyzing the specific metabolic changes of this disease, so as to conduct disease monitoring and efficacy evaluation.
Cerebrospinal fluid (CSF) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  The cerebrospinal fluid was examined by means of biochemical, transcriptomic, epigenetic and other methods.
Fugl-Meyer assessment scale (FMA) | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  The Fugl-Meyer Assessment (FMA) is a method used to evaluate the motor function status of patients of various ages. It is applicable in both clinical settings and research to determine the severity of diseases, describe motor recovery, and formulate plans as well as evaluate treatments.
Cranial MRI | Preoperative stage; One week after surgery; One week after device activation; Four weeks after device activation; Four weeks after discharge from hospital; Six months after discharge from hospital
  Utilize 3T and 7T magnetic resonance imaging to examine the resting state, occipital radiation spectroscopy, quantitative susceptibility mapping (QSM), and subvoxel imaging of the enrolled patients.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing TianTan Hospital, Beijing, Beijing Municipality
  - The 958 Hospital of Chinese People's Liberation Army, The Jiangbei Campus of Southwest Hospital, The First Affiliated Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - the Southwest hospital, Chongqing, Chongqing Municipality
  - Jingmen No.1 People's Hospital, Jingmen, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shanthanna H, Eldabe S, Provenzano DA, Bouche B, Buchser E, Chadwick R, Doshi TL, Duarte R, Hunt C, Huygen FJPM, Knight J, Kohan L, North R, Rosenow J, Winfree CJ, Narouze S. Evidence-based consensus guidelines on patient selection and trial stimulation for spinal cord stimulation therapy for chronic non-cancer pain. Reg Anesth Pain Med. 2023 Jun;48(6):273-287. doi: 10.1136/rapm-2022-104097. Epub 2023 Mar 30. PMID 37001888
- [Background] North R, Shipley J, Prager J, Barolat G, Barulich M, Bedder M, Calodney A, Daniels A, Deer T, DeLeon O, Drees S, Fautdch M, Fehrenbach W, Hernandez J, Kloth D, Krames ES, Lubenow T, North R, Osenbach R, Panchal SJ, Sitzman T, Staats P, Tremmel J, Wetzel T, American Academy of Pain Medicine. Practice parameters for the use of spinal cord stimulation in the treatment of chronic neuropathic pain. Pain Med. 2007 Dec;8 Suppl 4:S200-75. doi: 10.1111/j.1526-4637.2007.00388.x. No abstract available. PMID 17995571
- [Background] Powell MP, Verma N, Sorensen E, Carranza E, Boos A, Fields DP, Roy S, Ensel S, Barra B, Balzer J, Goldsmith J, Friedlander RM, Wittenberg GF, Fisher LE, Krakauer JW, Gerszten PC, Pirondini E, Weber DJ, Capogrosso M. Epidural stimulation of the cervical spinal cord for post-stroke upper-limb paresis. Nat Med. 2023 Mar;29(3):689-699. doi: 10.1038/s41591-022-02202-6. Epub 2023 Feb 20. PMID 36807682
- [Background] Kandhari S, Sharma D, Samuel S, Sharma G, Majumdar P, Edgerton VR, Gad P. Epidural Spinal Stimulation Enables Global Sensorimotor and Autonomic Function Recovery After Complete Paralysis: 1st Study From India. IEEE Trans Neural Syst Rehabil Eng. 2022;30:2052-2059. doi: 10.1109/TNSRE.2022.3158393. Epub 2022 Jul 27. PMID 35271446
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Luo S, Xu H, Zuo Y, Liu X, All AH. A Review of Functional Electrical Stimulation Treatment in Spinal Cord Injury. Neuromolecular Med. 2020 Dec;22(4):447-463. doi: 10.1007/s12017-019-08589-9. Epub 2020 Jan 8. PMID 31916220
- [Background] Moraud EM, Capogrosso M, Formento E, Wenger N, DiGiovanna J, Courtine G, Micera S. Mechanisms Underlying the Neuromodulation of Spinal Circuits for Correcting Gait and Balance Deficits after Spinal Cord Injury. Neuron. 2016 Feb 17;89(4):814-28. doi: 10.1016/j.neuron.2016.01.009. Epub 2016 Feb 4. PMID 26853304
- [Background] Rock AK, Truong H, Park YL, Pilitsis JG. Spinal Cord Stimulation. Neurosurg Clin N Am. 2019 Apr;30(2):169-194. doi: 10.1016/j.nec.2018.12.003. Epub 2019 Feb 18. PMID 30898269
- [Background] Dooley DM, Sharkey J, Keller W, Kasprak M. Treatment of demyelinating and degenerative diseases by electro stimulation of the spinal cord. Med Prog Technol. 1978 Nov 13;6(1):1-14. PMID 310508
- [Background] Shealy CN, Mortimer JT, Reswick JB. Electrical inhibition of pain by stimulation of the dorsal columns: preliminary clinical report. Anesth Analg. 1967 Jul-Aug;46(4):489-91. No abstract available. PMID 4952225
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Ni Y, Liu C, Tan L. Male Carrier of X-Linked Adrenal Leukodystrophy Due to 47, XXY Karyotype. JAMA Neurol. 2024 May 1;81(5):549-550. doi: 10.1001/jamaneurol.2024.0061. PMID 38436991
- [Background] Ombrone D, Giocaliere E, Forni G, Malvagia S, la Marca G. Expanded newborn screening by mass spectrometry: New tests, future perspectives. Mass Spectrom Rev. 2016 Jan-Feb;35(1):71-84. doi: 10.1002/mas.21463. Epub 2015 May 7. PMID 25952022
- [Background] van Egmond ME, Pouwels PJ, Boelens JJ, Lindemans CA, Barkhof F, Steenwijk MD, van Hasselt PM, van der Knaap MS, Wolf NI. Improvement of white matter changes on neuroimaging modalities after stem cell transplant in metachromatic leukodystrophy. JAMA Neurol. 2013 Jun;70(6):779-82. doi: 10.1001/jamaneurol.2013.629. PMID 23608771
- [Background] Matthes F, Stroobants S, Gerlach D, Wohlenberg C, Wessig C, Fogh J, Gieselmann V, Eckhardt M, D'Hooge R, Matzner U. Efficacy of enzyme replacement therapy in an aggravated mouse model of metachromatic leukodystrophy declines with age. Hum Mol Genet. 2012 Jun 1;21(11):2599-609. doi: 10.1093/hmg/dds086. Epub 2012 Mar 2. PMID 22388935
- [Background] Matzner U, Herbst E, Hedayati KK, Lullmann-Rauch R, Wessig C, Schroder S, Eistrup C, Moller C, Fogh J, Gieselmann V. Enzyme replacement improves nervous system pathology and function in a mouse model for metachromatic leukodystrophy. Hum Mol Genet. 2005 May 1;14(9):1139-52. doi: 10.1093/hmg/ddi126. Epub 2005 Mar 16. PMID 15772092
- [Background] Rosenberg JB, Kaminsky SM, Aubourg P, Crystal RG, Sondhi D. Gene therapy for metachromatic leukodystrophy. J Neurosci Res. 2016 Nov;94(11):1169-79. doi: 10.1002/jnr.23792. PMID 27638601
- [Background] Keller JL, Wang JI, Kang JY, Hanson JA, Kamath P, Swain JO, Raymond GV, Zackowski KM. Strength: a relevant link to functional performance in the neurodegenerative disease of adrenomyeloneuropathy. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1080-8. doi: 10.1177/1545968312441682. Epub 2012 Apr 27. PMID 22544816
- [Background] Moser HW, Moser AB, Naidu S, Bergin A. Clinical aspects of adrenoleukodystrophy and adrenomyeloneuropathy. Dev Neurosci. 1991;13(4-5):254-61. doi: 10.1159/000112170. PMID 1817030
- [Background] Moser HW, Mahmood A, Raymond GV. X-linked adrenoleukodystrophy. Nat Clin Pract Neurol. 2007 Mar;3(3):140-51. doi: 10.1038/ncpneuro0421. PMID 17342190
- [Background] Engelen M, Kemp S, Poll-The BT. X-linked adrenoleukodystrophy: pathogenesis and treatment. Curr Neurol Neurosci Rep. 2014 Oct;14(10):486. doi: 10.1007/s11910-014-0486-0. PMID 25115486
- [Background] Parikh S, Bernard G, Leventer RJ, van der Knaap MS, van Hove J, Pizzino A, McNeill NH, Helman G, Simons C, Schmidt JL, Rizzo WB, Patterson MC, Taft RJ, Vanderver A; GLIA Consortium. A clinical approach to the diagnosis of patients with leukodystrophies and genetic leukoencephelopathies. Mol Genet Metab. 2015 Apr;114(4):501-515. doi: 10.1016/j.ymgme.2014.12.434. Epub 2014 Dec 29. PMID 25655951